CLINICAL TRIAL: NCT06381180
Title: Wayne Warrior CAnnabis Research and Education: Cannabis and Behavioral Health
Brief Title: Warrior CARE: Cannabis Behavioral Health
Acronym: CBH
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Leslie Lundahl, Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Warrior CARE: CBH
Record Dates: First submitted 2023-01-17; First posted 2024-04-24 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Post Traumatic Stress Disorder; Cannabis Use; Suicide; Veterans; Marijuana
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Suicide; Marijuana Abuse | interventions — Dronabinol; Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- THC Group (Experimental): Cannabis with 5 mg THC; up to a maximum of 5 doses/day (max dose = 25 mg THC)
  Interventions: Drug: Tetrahydrocannabinol
- CBD Group (Experimental): Cannabis with 5 mg CBD; up to a maximum of 5 doses/day (max dose = 25 mg CBD)
  Interventions: Drug: Cannabidiol
- THC & CBD Group (Experimental): Cannabis with 5 mg THC and 5 mg CBD; up to a maximum of 5 doses/day (max doses = 25 mg THC and 25 mg CBD)
  Interventions: Drug: Tetrahydrocannabinol; Drug: Cannabidiol
- Placebo Group (Active Comparator): Cannabis with <1mg THC and <1mg CBD; up to a maximum of 5 doses/day (max dose = <5 mg THC and <5 mg CBD)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tetrahydrocannabinol — Plant cannabis that will be smoked
  Other Names: THC
  Arms: THC & CBD Group; THC Group
Drug: Cannabidiol — Plant cannabidiol that will be smoked
  Other Names: CBD
  Arms: CBD Group; THC & CBD Group
Drug: Placebo — Plant will be smoked.
  Arms: Placebo Group

SUMMARY:
This study is a randomized, controlled clinical trial to examine the therapeutic potential of cannabinoids for treating veterans with PTSD and suicidal ideation.

DETAILED DESCRIPTION:
In this clinical trial, we will recruit veterans with PTSD who report using cannabis or have interest in trying cannabis for symptom relief. Veterans will be randomized into one of four different groups: THC (∆9-tetrahydrocannabinol), CBD (cannabidiol), THC+CBD, and Placebo, and undergo a 12-week treatment phase where they will be asked to smoke their assigned cannabis dose every day for 12 weeks. Participants will complete weekly questionnaires regarding their mood, behavior and drug consumption. Furthermore, there is a laboratory component that will assess cognition, fear conditioning, and other PTSD-related measures.

ELIGIBILITY:
Inclusion Criteria:

* a healthy veteran who has served in a branch of the US armed forces
* report using cannabis within the past year
* currently meet DSM-5 criteria for PTSD and a score of 25 or greater on the CAPS-5 (the anchor, or index, trauma does not have to be related to military service)
* between the ages of 19-69 years old
* not seeking treatment for Cannabis Use Disorder
* stable (i.e., under the care of a physician or therapist and not experiencing acute symptoms) on psychotropic medications and/or psychotherapy before the study begins (participants can be in treatment for PTSD)
* agree to adhere to study procedures

Exclusion Criteria:

* pregnant, lactating, or heterosexually active women and not using medically approved birth control
* current or past bipolar or psychotic disorder as determined using the SCID-5
* at immediate high risk for suicide based on the C-SSRS
* current SUD other than Nicotine Use Disorder and Alcohol Use Disorder (mild or moderate)
* allergies and/or other contradictions for using cannabis
* any clinically significant medical problems
* systolic/diastolic BP >140/90 mmHg or systolic BP <95 mmHg
* elevated liver function tests
* exhibit cognitive impairment (<80 IQ)
* enrolled in another clinical trial or have received any drug as part of a research study within 30 days of dosing
* used a prescription medication (with the exception of birth control) within 14 days of study entry that in the opinion of the medically responsible investigator will interfere with the safety of the participant or the study results
* unable to provide informed consent

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-09-22 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessing change in PTSD diagnosis and its symptom severity from pre-treatment to post-treatment using the CAPS-5 assessment. | Administered at a pre-treatment visit (at the initial screening visit); and at the four post-treatment visits (one week post-treatment and 3-, 6-, and 9-months post-treatment visits).
  PTSD diagnosis will be assessed using the Clinician-Administered PTSD Scale (CAPS-5) for DSM-5 Total Severity Score, a well-validated, semi-structured clinician interview that determines the presence and severity of PTSD symptoms and diagnosis consistent with the DSM-5 and allows for assessing changes in symptom severity over time.
Assessing change in PTSD diagnosis and its symptom severity throughout the study using the PCL-5 assessment | Administered at every study visit: both pre-treatment visits (the initial screening and baseline visit); during the 12-week treatment phase (all twelve weekly visits); and the four post-treatment visits (one week post-treatment and 3-, 6-, and 9-months
  The PCL-5 is a 20-item self-report measure that assesses DSM-5 symptoms of PTSD. The PCL-5 is used to monitor symptom change during and after treatment, screen individuals for PTSD, and make a provisional PTSD diagnosis. This assessment will also be used as a safety measure at all visits by assessing PTSD symptom severity.
Assessing Suicidality over time using the C-SSRS assessment. | Administered at a pre-treatment visit (at the initial screening visit); and at the four post-treatment visits (one week post-treatment and 3-, 6-, and 9-months post-treatment visits).
  The Columbia Suicide Severity Rating Scale (C-SSRS) is a clinician-administered interview assessing suicidal thoughts and behaviors over time. A baseline form is used to assess lifetime suicidal ideation, intensity, and behavior, and can be compared to current suicidal ideation and intensity assessed over the clinical trial.
Assessing Suicidality throughout the study using the SBQ-R assessment. | Administered at every study visit: both pre-treatment visits (the initial screening and baseline visit); during the 12-week treatment phase (all twelve weekly visits); and the four post-treatment visits (one week post-treatment and 3-, 6-, and 9-months
  The Suicide Behavior Questionnaire-Revised (SBQ-R) is a brief (4-item), self-administered questionnaire that taps into four dimensions of suicidality (lifetime ideation/attempt, frequency of recent ideation, risk of suicide attempt and self-reported likelihood of future suicidal behavior). This assessment will also be used as a safety measure at all visits by assessing suicidality.
Assessing mood and anxiety symptoms throughout the study using the BDI-II and STAI-Y Questionnaires. | Administered at every study visit: both pre-treatment visits (the initial screening and baseline visit); during the 12-week treatment phase (all twelve weekly visits); and the four post-treatment visits (one week post-treatment and 3-, 6-, and 9-months
  The Beck Depression Inventory-II (BDI-II) is a self-report depression checklist which assesses neurovegetative depressive symptoms. One item asks specifically about suicidal thoughts and will also be checked at every study visit as a safety measure. The State Trait Anxiety Inventory-Form Y (STAI-Y) is a 40-item questionnaire with two scales assessing state and trait anxiety (somatic and cognitive symptoms).

SECONDARY OUTCOMES:
Assess emotional state pre- and post-treatment using the PANAS questionnaire. | Administered at a pre-treatment visit (at the baseline visit); and at the first post-treatment visit (one week post-treatment).
  The Positive and Negative Affect Schedule (PANAS) is a 20-item self-report questionnaire, widely used measure of emotional state, which has excellent psychometric properties.
Assess feelings of loneliness pre- and post-treatment using UCLA's 3-ILS assessment. | Administered at a pre-treatment visit (at the initial screening visit); and at the first post-treatment visit (one week post-treatment).
  The UCLA Three-Item Loneliness Scale (3-ILS) assesses social isolation and feelings of loneliness.
Assess dissociative symptoms pre- and post-treatment using the MDI and DSS assessments. | Administered at a pre-treatment visit (at the baseline visit); and at the four post-treatment visits (one week post-treatment, and 3-, 6-, and 9-months post-treatment).
  The Multiscale Dissociation Inventory (MDI) is a self-report questionnaire of dissociative symptomatology over the past month. The Dissociation Tension Scale (DSS) is a self-report measure of dissociative symptoms sensitive to weekly changes.
Assess drug effects, liking, and symptoms after cannabis administration using the SCERF and SES visual analog scales. | Administered after cannabis administration; therefore, administered at the baseline visit and electronically during the 12-week treatment phase (at all twelve weekly visits).
  The Subjective Cannabis Effects Rating Form (SCERF) will ask participants to complete a Visual Analog Scale (VAS) of "good drug effect," "bad drug effect," "strength of drug effect," liking," "sedated," and "desire to take again" and indicate whether they thought they received active drug or placebo. The Subjective Effects Scale (SES) VAS is a 33-item scale which includes the phrase "I feel…" followed by adjectives describing a mood (e.g., "anxious", "friendly," "down," etc.), a drug effect (e.g., "high," "stimulated", "a good drug effect") or a physical symptom (e.g., "hungry," "tired," "restless").
Assess demographics using a self-report assessment | Administered once at a pre-treatment visit, specifically at the initial screening visit.
  Participants will be asked to complete a personal history form to assess age, gender, sex, gender identity, marital status, race/ethnicity, education, employment status, and annual income.
Assess toxicant exposure commonly experienced during war using the KGWIC and BPE assessments. | Administered once at a pre-treatment visit, specifically at the baseline visit.
  The Kansas Gulf War Illness Criteria (KGWIC) and the Burn Pit Exposure (BPE) are self-report questionnaires that contain items on toxicants commonly experienced as well as burn pit exposure during war.
Assess smoking habits and history using the FTND assessment | Administered once at a pre-treatment visit, specifically at the baseline visit.
  Subjects who smoke cigarettes will also complete the Fagerstrom Test for Nicotine Dependence (FTND) survey to assess smoking history and habits.
Assess general health and history pre- and post-treatment using the SF-36 assessment. | Administered at a pre-treatment visit (the baseline visit); and at the four post-treatment visits (one week post-treatment and 3-, 6-, and 9-months post-treatment visits).
  The Short Form 36 (SF-36) is a brief measure of overall self-reported health that is associated with other objective health measures. Scores will be examined to assess change in general health outcomes over time.
Assess healthcare utilization throughout the study. | Administered at both pre-treatment visits (the initial screening and baseline visit); and at two post-treatment visits (one week post-treatment and 3-months post-treatment visits).
  The Healthcare Utilization (HU) survey will also assess the number of times participants utilize emergency room, urgent care, specialist, and general practitioner services.
Assess pain pre- and post-treatment using the BPI assessment. | Administered at a pre-treatment visit (the baseline visit); and at the four post-treatment visits (one week post-treatment and 3-, 6-, and 9-months post-treatment visits).
  The Brief Pain Inventory (BPI) asks participants to identify areas on their body causing pain and rate the severity.
Assess sleepiness pre- and post-treatment using the ESS questionnaire. | Administered at a pre-treatment visit (the baseline visit); and at the four post-treatment visits (one week post-treatment and 3-, 6-, and 9-months post-treatment visits).
  The Epworth Sleepiness Scale (ESS) is a self-report questionnaire that will be used to assess daytime sleepiness, which is indicative of sleep problems.
Assess overall quality of life pre- and post-treatment using the QOL questionnaire. | Administered at a pre-treatment visit (the baseline visit); and at the four post-treatment visits (one week post-treatment and 3-, 6-, and 9-months post-treatment visits).
  The Quality of Life (QOL) inventory assesses satisfaction in 17 life areas (work, health, recreation, goals, etc.) and will be used to assess the quality of life changes.
Assess substance use throughout the study using the TLFB assessment. | Administered at every study visit: both pre-treatment visits (the initial screening and baseline visit); during the 12-week treatment phase (all twelve weekly visits); and the four post-treatment visits (one week post-treatment and 3-, 6-, and 9-months
  The Timeline Follow-Back (TLFB) will be used to record the time of cannabis use and route of administration as well as any alcohol and other drug use.
Assess neurocognitive and executive function pre- and post-treatment using the WCST, WMS, CVLT, HMDD, WCS, IGT tasks | Administered at a pre-treatment visit (the baseline visit); and at the four post-treatment visits (one week post-treatment and 3-, 6-, and 9-months post-treatment visits).
  Working Memory will be assessed using the Wechsler Memory Scale (WMS) and the California Verbal Learning Test (CVLT). The Wisconsin Card Sort Task (WCST) assesses abstraction and the ability to shift or maintain cognitive set. The Hypothetical Monetary Delay Discounting (HMDD) and the Iowa Gambling Task (IGT) measure decision-making. Lastly, the Word Color Stroop (WCS) task assesses selective attention capacity and skills.
Assess physiological measures throughout the study as a safety check | Administered at every study visit: both pre-treatment visits (the initial screening and baseline visit); during the 12-week treatment phase (all twelve weekly visits); and the four post-treatment visits (one week post-treatment and 3-, 6-, and 9-months
  Physiological measures include blood pressure, heart rate, oxygen saturation, and skin temperature checks at all study visits
Assess biological samples for genetic markers associated with the endocannabinoid system and other biomarkers (e.g., cortisol) and measure THC and CBD. | Biological samples may be collected at a pre-treatment (at the baseline visit); during the 12-week treatment phase; and at the four post-treatment visits (one week post-treatment and 3-, 6-, and 9-months post-treatment visits)
  Biological measures include collection of urine, saliva, and blood. Saliva will be used to measure biomarkers like cortisol and test for endocannabinoid levels. Urine will be used to measure THC and CBD and their metabolites. Blood plasma will be used to measure plasma concentrations of endocannabinoids, cannabinoids, and PUFA metabolites.

CONTACTS AND LOCATIONS:
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Tashkin DP, Roth MD. Pulmonary effects of inhaled cannabis smoke. Am J Drug Alcohol Abuse. 2019;45(6):596-609. doi: 10.1080/00952990.2019.1627366. Epub 2019 Jul 12. PMID 31298945
- [Background] Huang YH, Zhang ZF, Tashkin DP, Feng B, Straif K, Hashibe M. An epidemiologic review of marijuana and cancer: an update. Cancer Epidemiol Biomarkers Prev. 2015 Jan;24(1):15-31. doi: 10.1158/1055-9965.EPI-14-1026. PMID 25587109
- [Background] Taylor DR, Fergusson DM, Milne BJ, Horwood LJ, Moffitt TE, Sears MR, Poulton R. A longitudinal study of the effects of tobacco and cannabis exposure on lung function in young adults. Addiction. 2002 Aug;97(8):1055-61. doi: 10.1046/j.1360-0443.2002.00169.x. PMID 12144608
- [Background] Tashkin DP, Simmons MS, Sherrill DL, Coulson AH. Heavy habitual marijuana smoking does not cause an accelerated decline in FEV1 with age. Am J Respir Crit Care Med. 1997 Jan;155(1):141-8. doi: 10.1164/ajrccm.155.1.9001303.
- [Background] Brauer RW, Dutcher JA, Vorus WS. Effects of prolonged simultaneous exposure of CD-1 mice to high pressures and inert gas narcosis. J Appl Physiol (1985). 1986 Dec;61(6):2129-35. doi: 10.1152/jappl.1986.61.6.2129. PMID 3804920
- [Background] Baldwin GC, Tashkin DP, Buckley DM, Park AN, Dubinett SM, Roth MD. Marijuana and cocaine impair alveolar macrophage function and cytokine production. Am J Respir Crit Care Med. 1997 Nov;156(5):1606-13. doi: 10.1164/ajrccm.156.5.9704146. PMID 9372683
- [Background] Tetrault JM, Crothers K, Moore BA, Mehra R, Concato J, Fiellin DA. Effects of marijuana smoking on pulmonary function and respiratory complications: a systematic review. Arch Intern Med. 2007 Feb 12;167(3):221-8. doi: 10.1001/archinte.167.3.221. PMID 17296876
- [Background] Tashkin DP, Fligiel S, Wu TC, Gong H Jr, Barbers RG, Coulson AH, Simmons MS, Beals TF. Effects of habitual use of marijuana and/or cocaine on the lung. NIDA Res Monogr. 1990;99:63-87. No abstract available. PMID 2267014
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Background] Russell D, Peplau LA, Ferguson ML. Developing a measure of loneliness. J Pers Assess. 1978 Jun;42(3):290-4. doi: 10.1207/s15327752jpa4203_11. PMID 660402
- [Background] Stiglmayr C, Schimke P, Wagner T, Braakmann D, Schweiger U, Sipos V, Fydrich T, Schmahl C, Ebner-Priemer U, Kleindienst N, Bischkopf J, Auckenthaler A, Kienast T. Development and psychometric characteristics of the Dissociation Tension Scale. J Pers Assess. 2010 May;92(3):269-77. doi: 10.1080/00223891003670232. PMID 20408027
- [Background] Briere, J. (2002). Multiscale Dissociation Inventory Professional Manual. Odessa, Florida: Psychological Assessment Resources.
- [Background] Delis DC, Freeland J, Kramer JH, Kaplan E. Integrating clinical assessment with cognitive neuroscience: construct validation of the California Verbal Learning Test. J Consult Clin Psychol. 1988 Feb;56(1):123-30. doi: 10.1037//0022-006x.56.1.123. No abstract available. PMID 3346437
- [Background] Budney AJ, Novy PL, Hughes JR. Marijuana withdrawal among adults seeking treatment for marijuana dependence. Addiction. 1999 Sep;94(9):1311-22. doi: 10.1046/j.1360-0443.1999.94913114.x. PMID 10615717
- [Background] Heishman SJ, Evans RJ, Singleton EG, Levin KH, Copersino ML, Gorelick DA. Reliability and validity of a short form of the Marijuana Craving Questionnaire. Drug Alcohol Depend. 2009 Jun 1;102(1-3):35-40. doi: 10.1016/j.drugalcdep.2008.12.010. Epub 2009 Feb 13. PMID 19217724
- [Background] Woskie SR, Bello A, Rennix C, Jiang L, Trivedi AN, Savitz DA. Burn Pit Exposure Assessment to Support a Cohort Study of US Veterans of the Wars in Iraq and Afghanistan. J Occup Environ Med. 2023 Jun 1;65(6):449-457. doi: 10.1097/JOM.0000000000002788. Epub 2023 Jan 11. PMID 36728333
- [Background] Steele L. Prevalence and patterns of Gulf War illness in Kansas veterans: association of symptoms with characteristics of person, place, and time of military service. Am J Epidemiol. 2000 Nov 15;152(10):992-1002. doi: 10.1093/aje/152.10.992. PMID 11092441
- [Background] Knopf, Alison. (2021). NIDA sets 5 mg of THC as standard cannabis unit for research. Alcoholism & Drug Abuse Weekly. 33. 6-7. 10.1002/adaw.33068.
- [Background] Lake S, Kerr T, Buxton J, Walsh Z, Marshall BD, Wood E, Milloy MJ. Does cannabis use modify the effect of post-traumatic stress disorder on severe depression and suicidal ideation? Evidence from a population-based cross-sectional study of Canadians. J Psychopharmacol. 2020 Feb;34(2):181-188. doi: 10.1177/0269881119882806. Epub 2019 Nov 5. PMID 31684805
- [Background] Kimbrel NA, Newins AR, Dedert EA, Van Voorhees EE, Elbogen EB, Naylor JC, Ryan Wagner H, Brancu M; VA Mid-Atlantic MIRECC Workgroup; Beckham JC, Calhoun PS. Cannabis use disorder and suicide attempts in Iraq/Afghanistan-era veterans. J Psychiatr Res. 2017 Jun;89:1-5. doi: 10.1016/j.jpsychires.2017.01.002. Epub 2017 Jan 5. PMID 28129565
- [Background] Americ, I.a.A.V.o. 2019 Member Survey. Perceptions and views of Iraq and Afghanistan veterans on the challenges and successes of the next greatest generation of veterans. . 2019; Available from: https://iava.org/iavas-2019-member-survey-results/.
- [Background] Olenick M, Flowers M, Diaz VJ. US veterans and their unique issues: enhancing health care professional awareness. Adv Med Educ Pract. 2015 Dec 1;6:635-9. doi: 10.2147/AMEP.S89479. eCollection 2015. PMID 26664252
- [Background] Boden MT, Babson KA, Vujanovic AA, Short NA, Bonn-Miller MO. Posttraumatic stress disorder and cannabis use characteristics among military veterans with cannabis dependence. Am J Addict. 2013 May-Jun;22(3):277-84. doi: 10.1111/j.1521-0391.2012.12018.x. PMID 23617872
- [Background] Adkisson K, Cunningham KC, Dedert EA, Dennis MF, Calhoun PS, Elbogen EB, Beckham JC, Kimbrel NA. Cannabis Use Disorder and Post-Deployment Suicide Attempts in Iraq/Afghanistan-Era Veterans. Arch Suicide Res. 2019 Oct-Dec;23(4):678-687. doi: 10.1080/13811118.2018.1488638. Epub 2018 Nov 17. PMID 29952737
- [Background] Hill MN, Bierer LM, Makotkine I, Golier JA, Galea S, McEwen BS, Hillard CJ, Yehuda R. Reductions in circulating endocannabinoid levels in individuals with post-traumatic stress disorder following exposure to the World Trade Center attacks. Psychoneuroendocrinology. 2013 Dec;38(12):2952-61. doi: 10.1016/j.psyneuen.2013.08.004. Epub 2013 Sep 10. PMID 24035186
- [Background] Hill MN, Miller GE, Ho WS, Gorzalka BB, Hillard CJ. Serum endocannabinoid content is altered in females with depressive disorders: a preliminary report. Pharmacopsychiatry. 2008 Mar;41(2):48-53. doi: 10.1055/s-2007-993211. PMID 18311684
- [Background] deRoon-Cassini TA, Stollenwerk TM, Beatka M, Hillard CJ. Meet Your Stress Management Professionals: The Endocannabinoids. Trends Mol Med. 2020 Oct;26(10):953-968. doi: 10.1016/j.molmed.2020.07.002. Epub 2020 Aug 28. PMID 32868170
- [Background] Abizaid A, Merali Z, Anisman H. Cannabis: A potential efficacious intervention for PTSD or simply snake oil? J Psychiatry Neurosci. 2019 Mar 1;44(2):75-78. doi: 10.1503/jpn.190021. No abstract available. PMID 30810022
- [Background] Zachary RA (1991) Shipley Institute of Living Scale: revised manual. Los Angeles: Western Psychological Services
- [Background] First MB, Williams JBW, Karg RS, Spitzer RL (2015) User's Guide for the Structured Clinical Interview for DSM-5 Disorders, Research Version (SCID-5-RV). Arlington, VA, American Psychiatric Association
- [Background] Weathers, F.W., et al., The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5). 2013, Washington DC: National Center for PTSD.
- [Background] Weathers, F.W., Litz, B.T., Keane, T.M., Palmieri, P.A., Marx, B.P., & Schnurr, P.P. (2013). The PTSD Checklist for DSM-5 (PCL-5). Scale available from the National Center for PTSD at www.ptsd.va.gov.
- [Background] Weathers FW, Bovin MJ, Lee DJ, Sloan DM, Schnurr PP, Kaloupek DG, Keane TM, Marx BP. The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5): Development and initial psychometric evaluation in military veterans. Psychol Assess. 2018 Mar;30(3):383-395. doi: 10.1037/pas0000486. Epub 2017 May 11. PMID 28493729
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Osman A, Bagge CL, Gutierrez PM, Konick LC, Kopper BA, Barrios FX. The Suicidal Behaviors Questionnaire-Revised (SBQ-R): validation with clinical and nonclinical samples. Assessment. 2001 Dec;8(4):443-54. doi: 10.1177/107319110100800409. PMID 11785588
- [Background] Beck, A.T., Steer, R.A., & Brown, G.K. (1996). Manual for the Beck Depression Inventory-II. San Antonio, TX: Psychological Corporation.
- [Background] Spielberger, C. D., Gorsuch, R. L., Lushene, R., Vagg, P. R., & Jacobs, G. A. (1983). Manual for the State-Trait Anxiety Inventory. Palo Alto, CA: Consulting Psychologists Press.
- [Background] Wechsler, D. (2009). Wechsler Memory Scale - 4th Edition. Pearson Assessments.
- [Background] BERG EA. A simple objective technique for measuring flexibility in thinking. J Gen Psychol. 1948 Jul;39:15-22. doi: 10.1080/00221309.1948.9918159. No abstract available. PMID 18889466
- [Background] Milner, B. (1963). Effects of different brain lesions on card sorting. Archives of Neurology, 9, 90-100.
- [Background] Bechara A, Damasio H, Tranel D, Damasio AR. Deciding advantageously before knowing the advantageous strategy. Science. 1997 Feb 28;275(5304):1293-5. doi: 10.1126/science.275.5304.1293. PMID 9036851
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Frisch, M.B., Cornell, J., Villanueva, M. & Retzlaff, P.J. (1992). Clinical validation of the quality of life inventory: A measure of life satisfaction for treatment planning and outcome assessment. Psychological Assessment, 4, 92-101.
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Marczylo TH, Lam PM, Nallendran V, Taylor AH, Konje JC. A solid-phase method for the extraction and measurement of anandamide from multiple human biomatrices. Anal Biochem. 2009 Jan 1;384(1):106-13. doi: 10.1016/j.ab.2008.08.040. Epub 2008 Sep 18. PMID 18823934
- [Background] Haney M, Ward AS, Comer SD, Foltin RW, Fischman MW. Abstinence symptoms following smoked marijuana in humans. Psychopharmacology (Berl). 1999 Feb;141(4):395-404. doi: 10.1007/s002130050849. PMID 10090647
- [Background] Haney M, Hart CL, Ward AS, Foltin RW. Nefazodone decreases anxiety during marijuana withdrawal in humans. Psychopharmacology (Berl). 2003 Jan;165(2):157-65. doi: 10.1007/s00213-002-1210-3. Epub 2002 Nov 19. PMID 12439626
- [Background] Bilgin M, Bindila L, Graessler J, Shevchenko A. Quantitative profiling of endocannabinoids in lipoproteins by LC-MS/MS. Anal Bioanal Chem. 2015 Jul;407(17):5125-31. doi: 10.1007/s00216-015-8559-8. Epub 2015 Mar 18. PMID 25782872
- [Background] Gachet MS, Rhyn P, Bosch OG, Quednow BB, Gertsch J. A quantitiative LC-MS/MS method for the measurement of arachidonic acid, prostanoids, endocannabinoids, N-acylethanolamines and steroids in human plasma. J Chromatogr B Analyt Technol Biomed Life Sci. 2015 Jan 22;976-977:6-18. doi: 10.1016/j.jchromb.2014.11.001. Epub 2014 Nov 18. PMID 25436483
- [Background] Marczylo TH, Lam PM, Amoako AA, Konje JC. Anandamide levels in human female reproductive tissues: solid-phase extraction and measurement by ultraperformance liquid chromatography tandem mass spectrometry. Anal Biochem. 2010 May 15;400(2):155-62. doi: 10.1016/j.ab.2009.12.025. Epub 2009 Dec 22. PMID 20026294
- [Background] Watkins BA, Kim J, Kenny A, Pedersen TL, Pappan KL, Newman JW. Circulating levels of endocannabinoids and oxylipins altered by dietary lipids in older women are likely associated with previously identified gene targets. Biochim Biophys Acta. 2016 Nov;1861(11):1693-1704. doi: 10.1016/j.bbalip.2016.07.007. Epub 2016 Jul 22. PMID 27452639
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865